CLINICAL TRIAL: NCT02472197
Title: Morcellator Versus Resectoscope in the Treatment of Uterine Polyps by Hysteroscopy
Acronym: RESMO
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Strasbourg, France (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 6043
Record Dates: First submitted 2015-06-05; First posted 2015-06-15 (Estimated); Last update posted 2025-12-19 (Actual); Status verified 2025-12

CONDITIONS: Endometrial Polyps
Keywords: Endometrial polyp; Hysteroscopic resection; Morcellation

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- morcellation (Experimental)
  Interventions: Procedure: Hysteroscopic morcellation
- standard resection (Active Comparator)
  Interventions: Procedure: Standard hysteroscopic resection

INTERVENTIONS:
Procedure: Hysteroscopic morcellation — The endometrial polyp is resected by a transcervical approach. During the procedure, the polyp is placed by suction against the window of the device, then cut by mechanical energy, in chips which are directly aspirated by the device.
  Arms: morcellation
Procedure: Standard hysteroscopic resection — The endometrial polyp is resected by a transcervical approach in several chips using a mono or bipolar cove after distension of the uterine cavity under endoscopic control.
  Arms: standard resection

SUMMARY:
Intrauterine pathologies are currently treated by hysteroscopic resection. In this surgical procedure, the intrauterine pathology is resected by a transcervical approach in several fragments using a mono or bipolar cove after distension of the uterine cavity and by endoscopic control. The main risks of this surgery are: uterine perforation and OHIA (operative hysteroscopy intravascular absorption) syndrome. Hysteroscopic morcellators are new intrauterine devices, recently appeared on the French market.

In comparison to classical resectors, morcellators have several theoretical advantages:

* A smaller instrument diameter with potentially a lower risk of uterine perforation and cervical laceration during the dilatation procedure,
* The use of physiological serum, eliminating the risk of neurological toxicity of glycine,
* The risk of electrical accident is canceled (internal or external burns due to leakage current),
* A decreased risk of air embolism, due to the absence of bubbles' production,
* The instrument is always under visual control, the perforation risk by the active instrument is therefore very limited,
* The vision is not obscured by the fragments or by the bubbles,
* The treatment of pre-ostial pathologies, not always easy in classical resections, could be facilitated,
* the absence of thermal effect, and therefore a potentially lower endometrial aggression, is interesting in women with reproductive desire,
* Absence of chips management, limiting the entry and exit movements in the uterine cavity, improving the vision, reducing the infectious and traumatic risks, specially uterine perforation and air embolism,
* Morcellation could preserve tissues for histological analysis of possible malignancy (compared to techniques using heat, coagulation, vaporization),
* Easy learning in comparison to the time-consuming learning of classical hysteroscopic resection,
* Generated additional cost could be partly amortized by reducing operating time and complications.

It seemed useful to study this new technology.

The primary purpose was to compare the time of hysteroscopic treatment of uterine polyps between a hysteroscopic morcellator the UNIDRIVE S III / DrillCut-X II-GYN-Shaver (Integrated Bigatti Shaver IBS), Storz®, and a conventional resectoscope.

The secondary purposes were to compare the efficiency, complications and comfort of these techniques.

ELIGIBILITY:
Inclusion Criteria:

* All major patients with single endometrial polyp,
* Confirmed by a diagnostic hysteroscopy
* Greater than or equal to one centimeter in size with no upper size limit
* Patient giving informed consent
* Subject belonging to a social security organisme

Exclusion Criteria:

* Ongoing pregnancy or breastfeeding
* Progressive malignant gynecological pathology
* Evolutionary Genital infection
* Suspected malignancy before surgery
* Multiple Polyps
* Polypoid hyperplasia
* Associated submucosal myoma
* Person under guardianship
* Patient with contraindication to general anesthesia or spinal anesthesia
* Person in an exclusion period (determined by a previous or ongoing study)
* Inability to give the eprosn informed information (comprehension difficulties ...)

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 90 (Actual)
Dates: Start 2015-09 (Actual); Primary Completion 2018-07 (Actual); Study Completion 2018-07 (Actual)

PRIMARY OUTCOMES:
Morcellation or resection time (minutes) | From the cervical dilatation just before introducing the operative device until removal of the operative device assessed up to 25 minutes

SECONDARY OUTCOMES:
The completeness of resection or not, | 10 weeks after surgery
The total operating time (in minutes): | from the beginning of diagnostic hysteroscopy to the end of operative hysteroscopy resection and removal of the operative device, assessed up to 25 minutes
The amount of serum used (mL) | At the end of surgery
Perioperative complications, | 10 weeks after surgery
The quality of vision defined by the operator on a scale of 0 to 5, | At the end of surgery
Persistence or not of the disease | 10 weeks after surgery
  evaluated by hysteroscopy
The occurrence of secondary adhesions | 10 weeks after surgery

CONTACTS AND LOCATIONS:
Overall Officials: Olivier GARBIN, MD, Principal Investigator — University Hospital, Strasbourg, France
Locations (1):
- University Hospital, Strasbourg, france, Strasbourg, France

REFERENCES:
- [Result] Stoll F, Lecointre L, Meyer N, Faller E, Host A, Hummel M, Boisrame T, Akladios C, Garbin O. Randomized Study Comparing a Reusable Morcellator with a Resectoscope in the Hysteroscopic Treatment of Uterine Polyps: The RESMO Study. J Minim Invasive Gynecol. 2021 Apr;28(4):801-810. doi: 10.1016/j.jmig.2020.07.007. Epub 2020 Jul 16. PMID 32681995